CLINICAL TRIAL: NCT06701539
Title: Effect of Nerve Block With Liposome Bupivacaine for Postoperative Pain After Craniotomy: A Randomized Control Trial
Brief Title: Liposomal Bupivacaine for Postoperative Pain After Craniotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Head of Anesthesiology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Libu20241120
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Liposome Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposome bupivacaine group (Experimental)
  Interventions: Drug: Liposome bupivacaine group
- Ropivacaine group (Active Comparator)
  Interventions: Drug: Ropivacaine group

INTERVENTIONS:
Drug: Liposome bupivacaine group — After standardized anesthesia induction, bilateral scalp nerve block (supprorbital nerve, auriculotemporal nerve, major occipital nerve, minor occipital nerve) was performed with liposome bupivacaine stock solution, and 1-2ml was injected into each block site.
  Arms: Liposome bupivacaine group
Drug: Ropivacaine group — After standardized anesthesia induction, bilateral scalp nerve block (supraorbital nerve, auriculotemporal nerve, major occipital nerve, minor occipital nerve) was administered with 0.5% ropivacaine, and 1-2ml was injected into each block site.
  Arms: Ropivacaine group

SUMMARY:
Acute postoperative pain is a common postoperative adverse reaction. It refers to acute pain that occurs immediately after surgery and usually lasts no longer than 3-7. Among the craniotomy approaches, patients undergoing supratentorial craniotomy with temporal approach had a higher incidence of moderate to severe pain within 24 hours. In the management of postoperative acute pain, multimodal analgesia is recommended. Liposomal bupivacaine was encapsulated by liposomal vesicles and released slowly, lasting up to 72 hours. The long action time also makes the time window of postoperative acute pain completely covered, thus helping patients better control pain. At present, there is an obvious lack of clinical studies on the effectiveness and specific duration of liposome bupivacaine for postoperative acute pain, especially in neurosurgical craniotomy population with transtemporal incision approach, which is a high-risk group for postoperative pain in neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old;
* Patients undergoing craniotomy tumor resection via frontotemporal approach, temporal base approach or temporal occipital approach;
* ASA grade I ~ III;
* Sign informed consent.

Exclusion Criteria:

* Previous history of combined drug allergy;
* Patients with a history of severe chronic pain;
* Long-term history of analgesic drug use;
* Patients with aphasia and other inability to cooperate with the scale were evaluated;
* Patients with mental system diseases;
* Patients with incomplete function of vital organs (heart, lung, liver, kidney);
* History of drug and drug abuse;
* BMI≥35kg/m2;
* Pregnant or lactating patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time of first incision pain within 72 hours after surgery | 72 hours after surgery